CLINICAL TRIAL: NCT07015437
Title: A Randomized, Controlled, Single-Blind, 2-Arm Parallel Study to Assess the Recovery and Lifespan of Radiolabeled Autologous INTERCEPT Red Blood Cells Prepared Using the INTERCEPT Blood System for RBCs With AS-1
Brief Title: A Recovery and Lifespan Study Using INTERCEPT Red Blood Cells Prepared Using the INTERCEPT Blood System for RBCs With AS-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CLI 00182
Record Dates: First submitted 2025-04-28; First posted 2025-06-11 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Healthy Subjects
Keywords: INTERCEPT; Red Blood Cells; RBC; Pathogen Inactivation; Pathogen reduction; Cerus; Survival; Radiolabel; Autologous; Recovery
MeSH Terms: interventions — Erythrocyte Count

STUDY DESIGN:
Who Masked: Participant
Masking Description: The subjects are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test RBCs will be prepared with the INTERCEPT Blood System for RBCs (Experimental): One unit of WB (500 ±50 mL) will be collected from subjects randomized to the Test treatment arm for preparation of the Test RBCs. The Test RBCs will be prepared with the INTERCEPT Blood System for RBCs with AS-1, within 24 hours or 25 to 48 hours post collection (depending on randomization assignment) and stored at 1°C to 6°C for 35 days. On Day 35 the subject will receive a single intravenous infusion of approximately 10 to 30 mL of Day 35 autologous 51Cr radiolabeled Test RBCs.
  Interventions: Device: INTERCEPT Blood System for RBCs; Other: Infusion of autologous radiolabeled RBCs
- Control RBC components will be prepared according to the site standard operating procedures (Experimental): One unit of WB (500 ±50 mL) will be collected from subjects randomized to the Control treatment arm for preparation of the Control RBCs in AS-1. The Control RBC components will be prepared and stored at 1°C to 6°C, according to the site standard operating procedures, for 35 days. On Day 35 the subject will receive a single intravenous infusion of approximately 10 to 30 mL of Day 35 51Cr autologous radiolabeled Control RBCs.
  Interventions: Other: Infusion of autologous radiolabeled RBCs

INTERVENTIONS:
Device: INTERCEPT Blood System for RBCs — RBCs treated with the INTERCEPT Blood System for RBCs
  Arms: Test RBCs will be prepared with the INTERCEPT Blood System for RBCs
Other: Infusion of autologous radiolabeled RBCs — Subject will receive a single intravenous infusion of approximately 10 to 30 mL of autologous Day 35 51Cr radiolabeled RBCs and fresh 99mTc RBCs.

SUMMARY:
The objective of this trial is to assess the post-infusion viability of INTERCEPT RBCs by measuring the 24-hour post-infusion recovery and lifespan of autologous RBCs prepared with the INTERCEPT Blood System for RBC with AS-1 after 35 days post collection storage in comparison to untreated AS-1 RBCs stored for 35 days.

DETAILED DESCRIPTION:
Study Design

This trial is designed as a prospective, randomized, controlled, single-blind (subject blinded), 2-arm parallel study to evaluate 24-hour post-infusion recovery and lifespan of 35-day-old autologous RBCs prepared with the INTERCEPT Blood System for RBCs with AS-1. Each subject will be infused with an aliquot of autologous radiolabeled INTERCEPT-treated (Test) or untreated (Control) AS-1 RBCs. During the study period each study subject will donate a whole blood (WB) component which will be processed to produce a leukocyte reduced AS-1 RBC component. Depending on the randomization assignment of the subject (Test or Control) the RBCs in AS-1 will be processed as a Test component (either within 24 hours or 25-48 hours of collection, depending on randomization) or Control component. On Day 35, an aliquot (10-30 mL) of study RBCs will be aseptically removed from the Test or Control RBC component and radiolabeled with 51Cr for assessment of recovery and lifespan.

On Day 35, the same healthy subjects will return to the site and provide a fresh sample of heparinized blood (approximately 10 mL), the fresh autologous RBCs from this sample will be radiolabeled with 99mTc for measurement of blood volume.

The 51Cr (Test or Control) and 99mTc (fresh RBCs) radiolabeled samples (approximately 10-30 mL) will be simultaneously infused into the subject. To measure RBC recovery and blood volume, subject blood samples will be collected at the following time points after completion of the infusion: approximately 5, 7.5, 10, 12.5, 15, 20, and 30 minutes (Day 35) and at 24 ±4 hours (Day 36). To measure the RBC lifespan post infusion, additional subject blood samples will be collected. 51Cr activity will be measured at approximately 48 hours (Day 37), 72 hours (Day 38), 7 days (Day 42) post-infusion, and then weekly through 35 days post-infusion (approximately Days 49, 56, 64, and 70) for Test and Control subjects. For Test subjects, as an additional measure of circulating INTERCEPT RBCs, the proportion of acridine positive RBCs and level of acridine on Test RBCs will be evaluated. Post-infusion RBC samples will be frozen at approximately 30 minutes on Day 35 and on Days 36, 37, 38, 42, 49, 56, 64, 70, and 90.

Subjects will be monitored for adverse events (serious and non-serious) for 24 hours following the WB donation and approximately 24 hours following infusion of study RBCs. Only serious and treatment emergent adverse events, including transfusion reactions, will be assessed at subsequent post-infusion visits.

Samples for in vitro RBC testing (see in vitro evaluation of RBCs below) will be collected from RBC components at input, post-INTERCEPT (Test only), and after 35 days of storage (Test and Control).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Complete blood count (CBC) and serum chemistry values within normal limits or outside of normal reference range but determined by the Investigator, and consultation with the Sponsor, to be not clinically significant.
* Meet FDA, AABB, or institutional guidelines for allogeneic WB donation, including viral marker testing, with the following exceptions:
* Meeting allogeneic deferral criteria due to travel, tattoos/piercings and male to male sexual contact would be acceptable, subject to the Investigator's discretion.
* Subjects of childbearing potential must agree to use a medically acceptable method of contraception throughout the study.
* Signed and dated informed consent form

Exclusion Criteria:

* History of RBC autoantibodies, autoimmune hemolytic anemia, RBC allo-antibodies, or other autoimmune disease
* History of congenital red cell disorders (including self-reported glucose 6 phosphate dehydrogenase (G- 6PD) deficiency, sickle cell trait and thalassemia minor trait)
* Positive DAT or IAT at study entry
* Immunosuppressive therapy (e.g., oral or IV prednisone) within the past 28 days
* Treatment with any medication known to affect RBC viability
* Pregnant or nursing females
* Participation in another interventional clinical study currently or has received an investigational drug within the past 28 days
* Less than three months from receiving an infusion of a radiolabeled blood component.
* Reenrollment in the same treatment group for which the subject previously contributed recovery and survival data in this study.
* Non study blood component donation throughout the study
* Preexisting antibody specific to INTERCEPT RBCs
* History of known hypersensitivity to chromium or technetium

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
The percentage of infused 35-day-old autologous 51Cr-labeled Test/INTERCEPT or Control RBCs remaining in circulation 24 hours post-infusion | Pre-transfusion and 5, 7.5, 10, 12.5, 15, 20, and 30 minutes and at 24 hours after infusion
  The 24-hour recovery will be calculated using the subject's blood volume derived from infusion of 99mTc-labeled fresh RBCs.

SECONDARY OUTCOMES:
. The percentage of infused 35-day-old autologous 51Cr-labeled Test/INTERCEPT or Control RBCs remaining in circulation 24 hours post-infusion | Pre-transfusion and 5, 7.5, 10, 12.5, 15, 20, and 30 minutes and at 24 hours after infusion
  The 24-hour recovery will be calculated using the subject's blood volume derived the subject's height and weight.
. The number of days 51Cr-labeled Test/INTERCEPT or Control RBCs remain in circulation up to post-infusion | Over 35 days post infusion
  The value will be derived by measurement of detectable 51Cr- labeled RBC with time
Hemolysis (<1%) | 35 days
  Proportion of RBC component hemolysis on Day 35 (<1%).

OTHER OUTCOMES:
Adverse Events | 90 days
  Incidence of treatment emergent adverse events possibly, probably, or definitely related to the study RBCs over the course of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - American Red Cross Research Laboratory, Norfolk, Virginia